CLINICAL TRIAL: NCT05652725
Title: Radicle™ Clarity: A Randomized, Blinded, Placebo-Controlled Direct-to-Consumer Study of Health and Wellness Products on Cognitive Function and Other Health Outcomes
Brief Title: Radicle Clarity: A Study of Health and Wellness Products on Mental Clarity and Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-2306
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Cognitive Function

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on gender at birth then randomized to one of the study arm
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Placebo Control 1 (Placebo Comparator): Clarity Product Form 1 - control
  Interventions: Dietary Supplement: Placebo Control Form 1
- Placebo Control 2 (Placebo Comparator): Clarity Product Form 2 - control
  Interventions: Dietary Supplement: Placebo Control Form 2
- Placebo Control 3 (Placebo Comparator): Clarity Product Form 3 - control
  Interventions: Dietary Supplement: Placebo Control Form 3
- Placebo Control 4 (Placebo Comparator): Clarity Product Form 4 - control
  Interventions: Dietary Supplement: Placebo Control Form 4
- Active Product 1.1 (Experimental): Clarity Product Form 1 - active product 1
  Interventions: Dietary Supplement: Clarity Active Study Product 1.1 Usage
- Active Product 2.1 (Experimental): Clarity Product Form 2 - active product 1
  Interventions: Dietary Supplement: Clarity Active Study Product 2.1 Usage
- Active Product 3.1 (Experimental): Clarity Product Form 3 - active product 1
  Interventions: Dietary Supplement: Clarity Active Study Product 3.1 Usage
- Active Product 4.1 (Experimental): Clarity Product Form 4 - active product 1
  Interventions: Dietary Supplement: Clarity Active Study Product 4.1 Usage
- Active Product 4.2 (Experimental): Clarity Product Form 4 - active product 2
  Interventions: Dietary Supplement: Clarity Active Study Product 4.2 Usage
- Active Product 4.3 (Experimental): Clarity Product Form 4 - active product 3
  Interventions: Dietary Supplement: Clarity Active Study Product 4.3 Usage
- Placebo Control 5 (Placebo Comparator): Clarity Product Form 5 - control
  Interventions: Dietary Supplement: Placebo Control Form 5
- Active Product 5.1 (Experimental): Clarity Product Form 5 - active product 1
  Interventions: Dietary Supplement: Clarity Active Study Product 5.1 Usage
- Active Product 5.2 (Experimental): Clarity Product Form 5 - active product 2
  Interventions: Dietary Supplement: Clarity Active Study Product 5.2 Usage

INTERVENTIONS:
Dietary Supplement: Clarity Active Study Product 1.1 Usage — Participants will use their Radicle Clarity Active Study Product 1.1 as directed for a period of 6 weeks.
  Arms: Active Product 1.1
Dietary Supplement: Clarity Active Study Product 2.1 Usage — Participants will use their Radicle Clarity Active Study Product 2.1 as directed for a period of 6 weeks.
  Arms: Active Product 2.1
Dietary Supplement: Clarity Active Study Product 3.1 Usage — Participants will use their Radicle Clarity Active Study Product 3.1 as directed for a period of 6 weeks.
  Arms: Active Product 3.1
Dietary Supplement: Clarity Active Study Product 4.1 Usage — Participants will use their Radicle Clarity Active Study Product 4.1 as directed for a period of 6 weeks.
  Arms: Active Product 4.1
Dietary Supplement: Clarity Active Study Product 4.2 Usage — Participants will use their Radicle Clarity Active Study Product 4.2 as directed for a period of 6 weeks.
  Arms: Active Product 4.2
Dietary Supplement: Clarity Active Study Product 4.3 Usage — Participants will use their Radicle Clarity Active Study Product 4.3 as directed for a period of 6 weeks.
  Arms: Active Product 4.3
Dietary Supplement: Placebo Control Form 1 — Participants will use their Placebo Control Form 1 as directed for a period of 6 weeks.
  Arms: Placebo Control 1
Dietary Supplement: Placebo Control Form 2 — Participants will use their Placebo Control Form 2 as directed for a period of 6 weeks.
  Arms: Placebo Control 2
Dietary Supplement: Placebo Control Form 3 — Participants will use their Placebo Control Form 3 as directed for a period of 6 weeks.
  Arms: Placebo Control 3
Dietary Supplement: Placebo Control Form 4 — Participants will use their Placebo Control Form 4 as directed for a period of 6 weeks.
  Arms: Placebo Control 4
Dietary Supplement: Placebo Control Form 5 — Participants will use their Placebo Control Form 5 as directed for a period of 6 weeks.
  Arms: Placebo Control 5
Dietary Supplement: Clarity Active Study Product 5.1 Usage — Participants will use their Radicle Clarity Active Study Product 5.1 as directed for a period of 6 weeks.
  Arms: Active Product 5.1
Dietary Supplement: Clarity Active Study Product 5.2 Usage — Participants will use their Radicle Clarity Active Study Product 5.2 as directed for a period of 6 weeks.
  Arms: Active Product 5.2

SUMMARY:
A randomized, blinded, placebo-controlled direct-to-consumer study of health and wellness products on mental clarity and other health outcomes

DETAILED DESCRIPTION:
This is a randomized, blinded, placebo-controlled study conducted with adult participants, age 21 and older and residing in the United States.

Eligible participants will (1) endorse a desire for better concentration, (2) indicate an interest in taking a health and wellness product to potentially help their concentration, and (3) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants with known liver or kidney disease, heavy drinkers, and those who report they are pregnant, trying to become pregnant, or breastfeeding will be excluded. Those taking certain medications will be excluded.

Self-reported data are collected electronically from eligible participants over 7 weeks. Participant reports of health indicators will be collected during baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 21 years of age and older at the time of electronic consent, inclusive of all ethnicities, races, genders and/or gender identities
* Resides in the United States
* Endorses better concentration as a primary desire
* Selects concentration and/or looking to improve their concentration as a reason for their interest in taking a health and wellness product
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

* Reports being pregnant, trying to become pregnant, or breastfeeding
* Unable to provide a valid US shipping address and mobile phone number
* The calculated validated health survey (PRO) score during enrollment represents less than mild impairment or severity
* Reports a diagnosis of liver or kidney disease
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Reports current enrollment in a clinical trial
* Lack of reliable daily access to the internet
* Reports current or recent (within 3 months) use of chemotherapy or immunotherapy
* Reports taking medications with a known moderate or severe interaction with any of the active ingredients studied or a substantial safety risk: Anticoagulants, a medication that warns against grapefruit consumption, corticosteroids at doses greater than 5 mgs per day, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, or MAOIs (monoamine oxidase inhibitors)
* Reports a diagnosis of heart disease when a known contraindication exists for any of the active ingredients studied: NYHA (New York Heart Association) Class III or IV congestive heart failure, Atrial fibrillation, Uncontrolled arrhythmias

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4826 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Change in cognition (mental clarity) | 6 weeks
  Mean difference in cognition score as assessed by Patient Reported Outcome Measurement System (PROMIS) Cognitive Function Short Form 8A (scale 8-40; where the higher scores correspond to greater cognitive function)

SECONDARY OUTCOMES:
Change in executive functioning | 6 weeks
  Mean difference in cognition score as assessed by Adult Executive Functioning Inventory (ADEXI) (scale 1-5; with higher scores corresponding to lower executive functioning)
Change in sleep quality | 6 weeks
  Mean difference in sleep quality score as assessed by PROMIS Sleep Disturbance 4A (scale 4-20; with higher scores corresponding to greater sleep disturbance)
Change in energy (fatigue) | 6 weeks
  Mean difference in energy score as assessed by PROMIS Fatigue 4A (scale 4-20; where higher scores correspond to more severe fatigue)
Change in anxiety | 6 weeks
  Mean difference in anxiety score as assessed by PROMIS Anxiety 4A (scale 4-20; with higher scores corresponding to more severe anxiety)
Change in mood (emotional distress) | 6 weeks
  Mean difference in mood score as assessed by PROMIS Depression 4A (scale 4-20; where higher scores correspond to more severe depression)
Change in libido | 6 weeks
  Mean difference in libido score as assessed by PROMIS Sexual Interest 2.0 (scale 2-10; where higher scores correspond to greater sexual interest)
Minimal clinical importance difference (MCID) in cognitive function | 6 weeks
  Likelihood of achieving a MCID in cognitive function, as measured by PROMIS Cognitive Function Short Form 8A (scale 8-40; where the higher scores correspond to greater cognitive function)

CONTACTS AND LOCATIONS:
Overall Officials: Emily K. Pauli, PharmD, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com